CLINICAL TRIAL: NCT00439166
Title: Effects of Treatment With Doxycycline and Rifampicin on Biomarkers of Alzheimer's Disease in the Cerebrospinal Fluid
Brief Title: Effects of Doxycycline and Rifampicin on Biomarkers of Alzheimer's Disease in the Cerebrospinal Fluid
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Sponsor
Organization: McMaster University (Other)
Allocation: Non-Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PSI 06-47
Record Dates: First submitted 2007-02-20; First posted 2007-02-23 (Estimated); Last update posted 2018-03-19 (Actual); Status verified 2017-03

CONDITIONS: Alzheimer's Disease
Keywords: doxycycline; rifampicin; cerebrospinal fluid; biomarkers; beta amyloid; tau
MeSH Terms: conditions — Alzheimer Disease; Plaque, Amyloid; Pick Disease of the Brain | interventions — Doxycycline; Rifampin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 AD combined doxycycline + rifampin (Experimental): Doxycycline 100 mg b.i.d. plus rifampin 300 mg o.d. for 12 months.
  Interventions: Drug: doxycycline; Drug: rifampicin
- 2 AD Doxycycline only (Experimental): Doxycycline 100 mg b.i.d. plus placebo matched to rifampin o.d. for 12 months.
  Interventions: Drug: doxycycline; Drug: Placebo matched to Rifampin
- 3 Rifampin only (Experimental): Rifampin 300 mg o.d. plus placebo matched to doxycycline b.i.d. for 12 months.
  Interventions: Drug: rifampicin; Drug: Placebo matched to doxycycline
- 4 Double Placebo (Placebo Comparator): Placebo matched to Doxycycline b.i.d. plus placebo matched to rifampin o.d. for 12 months.
  Interventions: Drug: Placebo matched to doxycycline; Drug: Placebo matched to Rifampin

INTERVENTIONS:
Drug: doxycycline — capsule, 100 mg, b.i.d., daily for 1 year
  Arms: 1 AD combined doxycycline + rifampin; 2 AD Doxycycline only
Drug: rifampicin — capsule, 300mg, o.d., daily for 11 months (administration starts in 2nd month of trial)
  Other Names: Rofact; Rifadin
  Arms: 1 AD combined doxycycline + rifampin; 3 Rifampin only
Drug: Placebo matched to doxycycline — Doxycycline-matched - blue capsule, b.i.d.,daily for 12 months
  Arms: 3 Rifampin only; 4 Double Placebo
Drug: Placebo matched to Rifampin — Rifampin-matched - red capsule, o.d., daily for 11 months starting at month 2.
  Arms: 2 AD Doxycycline only; 4 Double Placebo

SUMMARY:
This study will determine if biomarkers found in the cerebrospinal fluid of people with Alzheimer's disease, are affected by treatment with two common antibiotics, doxycycline and rifampicin, suggesting a disease-modifying effect of those treatments.

DETAILED DESCRIPTION:
Diagnostic markers in the cerebrospinal fluid (CSF) have become a rapidly growing research field. Potential disease-modifying drugs like the antibiotics rifampicin and doxycycline, highlight the need of improved diagnostic accuracy and offer the potential to examine how these treatments may actually exert their clinical effects.

Cerebrospinal fluid biomarkers (the 42 amino acid form of β-amyloid (Aβ), total tau, and phosphorylated tau) have been evaluated in scientific studies. Tau proteins are considered "state" markers, whereas Aβ(1-42) proteins can be used as "stage" markers. These CSF markers have high sensitivity to differentiate early AD from normal aging, depression, alcohol dementia and Parkinson's disease. When these biomarkers are used in combination with a medical history, clinical examination, laboratory tests and brain imaging, the diagnostic accuracy is improved.

Matrix metalloproteinase (MMP) dysregulation is thought to contribute to a variety of pathological conditions such as arthritis, cancer, atherosclerosis, aneurysms, nephritis, tissue ulcers, and fibrosis. In addition, MMP involvement has been demonstrated in the pathogenesis of a variety of CNS disorders, including bacterial and viral disorders, stroke, multiple sclerosis, ALS, and AD.

There is an inflammatory response in AD. This includes complement activation, elevated C-reactive protein (CRP), elevated pro-inflammatory cytokines (including IL-1-β, IL-6, TNF-α, TGF-β, S100-β), chemokine alterations (IL-8, MIP-1-α, MIP-1-β, MCP-1), and microglial.

We are measuring the biochemical markers of Aβ(1-40) and Aβ(1-42), P-tau and T-tau, matrix metalloproteinases (MMP-2, MMP-9), pro-inflammatory cytokines (IL-1beta, TNF-alpha), and anti-inflammatory cytokines (IL-4 and IL-10) at the start and one year after treatment in the multi-centered, randomized, controlled, trial of disease-modifying drugs rifampicin and/or and doxycycline to slow the progress of Alzheimer's disease by affecting the production of these biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age greater than or equal to 50 years
* Diagnosis of probable Alzheimer's disease by NINCDS-ADRDA criteria
* Standardized Mini-Mental State Examination score 14-26 inclusive
* A caregiver who consents to monitor study medications, report on patient function, bring the patient to visits, etc.
* Vision, hearing, language ability sufficient to complete standardized testing in English.
* Patient consents (or legal representative consents for patient)
* Generally stable level of health where patient may be reasonably expected to complete a 1 year trial

Exclusion Criteria:

* Other neurodegenerative diseases such as Lewy body or Parkinson's
* Cognitive impairment due to: acute trauma, subdural hematoma, hypoxic cerebral damage, B12 deficiency, infections such as AIDS or meningitis, cerebral neoplasia, endocrine deficiencies, mental retardation
* Significant cerebrovascular disease or multi-infarct dementia
* Intra-cranial pathology such as tumour
* Co-existing medical conditions such as epilepsy, major psychiatric conditions, depression (Cornell Depression in Dementia Scale score of 12 or more), significant liver, kidney, lung, metabolic or endocrine diseases
* Clinically significant cardiac disease such as uncontrolled angina or hypertension
* Anti-dementia treatments other than donepezil, galantamine, rivastigmine, memantine
* Enrollment in trials with other investigational drugs
* Antibiotic use more than one month in the last six months
* Allergy to doxycycline or rifampicin

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-02; Primary Completion 2010-04 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Clinical Dementia Rating scale | 12 months
Standardized Alzheimer's disease Assessment Scale -cognitive subscale | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: William Molloy, MB, FRCPC, Study Chair — McMaster University; Tricia KW Woo, MD, FRCPC, Principal Investigator — McMaster University; David D Cowan, MD, FRCPC, Principal Investigator — McMaster University; Brandon M Kucher, PhD, Principal Investigator — McMaster University; Alwin Cunje, MD, PhD, Principal Investigator — University of Ottawa; Tim I Standish, MA, Principal Investigator — McMaster University
Locations (1):
- St.Peter's Hospital, Hamilton, Ontario, Canada